CLINICAL TRIAL: NCT02406651
Title: A Phase IIa Study of Recombinant Human Interleukin-22 IgG2-Fc (F 652) in Combination With Systemic Corticosteroids for the Treatment of Newly Diagnosed Grade II-IV Lower Gastrointestinal Acute Graft-versus-Host Disease (aGVHD) in Hematopoietic Stem Cell Transplantation Recipients (HSCT)
Brief Title: Study of IL-22 IgG2-Fc (F-652) for Subjects With Grade II-IV Lower GI aGVHD
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: EVIVE Biotechnology (Industry)
Collaborators: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GC-652-02
Record Dates: First submitted 2015-03-19; First posted 2015-04-02 (Estimated); Results first posted 2021-07-22 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Acute Graft vs Host Disease
MeSH Terms: interventions — eflepedocokin alfa; Interleukin-22

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- F-652 and systemic coritcosteroids (Experimental): Subjects will be dosed once a week for four weeks with Recombinant Human Interleukin-22 IgG2-Fc (F-652). Dosing will be concurrent with systemic corticosteroids.
  Interventions: Drug: Recombinant Human Interleukin-22 IgG2-Fc (F-652); Drug: Systemic Corticosteroids

INTERVENTIONS:
Drug: Recombinant Human Interleukin-22 IgG2-Fc (F-652) — IV infusion of reconstitution lyophilized F-652.
  Other Names: IL-22
Drug: Systemic Corticosteroids — Prednisone (or equivalent) at the time of the onset of clinical symptoms consistent with GI and/or liver aGVHD, as per the standard of care. Prednisone (or equivalent) will be given at a dose of 2 mg/kg/day and tapered as needed.

SUMMARY:
A Phase IIa single arm open-label study to investigate the safety, tolerability, and PK of F-652 in combination with systemic corticosteroids in subjects who have undergone Hematopoietic Stem Cell Transplantation (HSCT) and have newly diagnosed grade II-IV lower GI acute Graft Verses Host Disease (aGVHD). Treatment with F-652 will be once a week for 4 weeks, with post treatment follow up visits on days 28, 56, 180 and 365.

DETAILED DESCRIPTION:
This is a Phase IIa single arm open-label study to investigate the safety, tolerability, and PK of F-652 in combination with systemic corticosteroids in subjects who have undergone HSCT and have newly diagnosed grade II-IV lower GI aGVHD. The HSCT may be derived from bone marrow, peripheral blood stem cells, or cord blood. The PK of F-652 in this subject population will be investigated. Subjects may be replaced if subject withdrawal is not related to safety or treatment response.

F-652 will be administered in conjunction with prednisone (or equivalent) at the time of the onset of clinical symptoms consistent with GI and/or liver aGVHD. Prednisone (or equivalent) will be given at a dose of 2 mg/kg/day and tapered as per protocol.

F-652 will be administered intravenously at a rate of 100 mL/hour for one hour once per week for four weeks. A total of 4 doses will be administered at a dose of 45 μg/kg each. Subjects will be followed for safety and efficacy through Day 180, and subject survival status will be collected at Day 365.

In the first stage of the trial, a total of 16 subjects will be enrolled. If six or fewer have a Day 28 treatment response, the trial will close due to a lack of efficacy. If seven or more have a response, an additional 11 subjects will be enrolled into study for a total sample size of 27. During the course of a subject's therapy, dose reduction may occur on an individual basis as per protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years and ≤80.
2. Newly diagnosed lower GI grade II-IV aGVHD with clinical diagnosis based on modified Keystone criteria1 following allogeneic HSCT using bone marrow, peripheral blood stem cells, or cord blood. Grading of aGVHD will be based on International Bone Marrow Transplant Registry (IBMTR) criteria.
3. Subjects are willing to undergo a biopsy to confirm lower GI aGVHD. Biopsy results are not needed to initiate treatment. However, if aGVHD is not confirmed histologically, treatment with F-652 will be discontinued.
4. Female subjects of childbearing potential who agree to practice 2 effective methods of contraception.
5. Male subjects, even if surgically sterilized (i.e. Status post-vasectomy) must agree to agree to practice contraception.
6. Have adequate renal function (Serum creatinine <3 mg/dL).
7. ANC >500/mm3.
8. Show evidence of a personally signed and dated informed consent document indicating that the subject (or legally acceptable representative) has been informed of all pertinent aspects of the trial.

Exclusion Criteria:

Subjects who met any of the following criteria were excluded from the study:

1. Evidence of relapse or progression of hematologic malignancy at the time of study enrollment.
2. Active uncontrolled infection. Subjects with a controlled infection receiving definitive therapy for 48 hours prior to enrollment were eligible.
3. Subjects requiring vasopressors or mechanical ventilation.
4. Subjects who had received previous systemic corticosteroids for the treatment of acute GI GVHD for longer than 5 days. Subjects who were treated with systemic corticosteroids for aGVHD for a prior allogeneic HSCT >12 months ago were eligible.
5. Subjects who received any corticosteroid therapy (for non-GVHD) at doses >0.5 mg/kg/day prednisone (or IV equivalent) within 7 days prior to the onset of GVHD therapy.
6. Subjects who developed aGVHD after unplanned donor lymphocyte infusion.
7. Subjects with chronic GVHD features (i.e., acute/chronic GVHD overlap syndrome or classical chronic GVHD).
8. History of psoriasis.
9. History of epithelial malignancies including melanoma or any carcinomas.
10. History or diagnosis of mantle cell lymphoma or anaplastic large cell lymphoma.
11. Subject was pregnant or breast-feeding.
12. Evidence of current uncontrolled cardiovascular conditions, including uncontrolled hypertension, uncontrolled cardiac arrhythmias, symptomatic congestive heart failure, unstable angina, or myocardial infarction within the past 6 months.
13. The subject or guardian was unable to give informed consent or unable to comply with the treatment protocol including appropriate supportive care, follow-up, and research tests.
14. The subject had tested positive for the Clostridium difficile (C. difficile) toxin within 7 days of study entry.
15. Cytotoxic, biologic, or investigational agents were not permitted throughout the study. These included, but were not limited to, ATG, alemtuzumab, rituximab, photopheresis, and thalidomide. Subjects who participated in any other investigational drug trial or had exposure to any other investigational agent, device, or procedure, within 4 weeks prior to screening and throughout the entire trial, except for trials of investigational drugs administered prophylactically for GVHD or CMV post-allogeneic HSCT. In this exception, the other investigational drug must have been discontinued upon enrolling (i.e., screening/sign ICF) into this study.
16. Any serious medical or psychiatric illness that could, in the Investigator's opinion, potentially have interfered with the completion of treatment according to this protocol.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-05-12 (Actual); Primary Completion 2019-04-09 (Actual); Study Completion 2020-03-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Doris Ponce, M.D., Principal Investigator — MSKCC
Locations (3):
- United States (3):
  - City of Hope, Duarte, California
  - MSKCC, New York, New York
  - MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Derived] Ponce DM, Alousi AM, Nakamura R, Slingerland J, Calafiore M, Sandhu KS, Barker JN, Devlin S, Shia J, Giralt S, Perales MA, Moore G, Fatmi S, Soto C, Gomes A, Giardina P, Marcello L, Yan X, Tang T, Dreyer K, Chen J, Daley WL, Peled JU, van den Brink MRM, Hanash AM. A phase 2 study of interleukin-22 and systemic corticosteroids as initial treatment for acute GVHD of the lower GI tract. Blood. 2023 Mar 23;141(12):1389-1401. doi: 10.1182/blood.2021015111. PMID 36399701

RESULTS

PARTICIPANT FLOW:
Groups:
- F-652 and Systemic Coritcosteroids: Subjects was dosed once a week for four weeks with Recombinant Human Interleukin-22 IgG2-Fc (F-652). Dosing was concurrent with systemic corticosteroids.
  Recombinant Human Interleukin-22 IgG2-Fc (F-652): IV infusion of reconstitution lyophilized F-652.
  Systemic Corticosteroids: Prednisone (or equivalent) was at the time of the onset of clinical symptoms consistent with GI and/or liver aGVHD, as per the standard of care. Prednisone (or equivalent) was given at a dose of 2 mg/kg/day and tapered as needed.
Period: Overall Study
Arm/Group | F-652 and Systemic Coritcosteroids
Started | 30
Completed | 27
Not Completed | 3
Not completed — 30 subjects dosed based on initial screening. 3 subjects were removed because they screened fail. | 3

BASELINE CHARACTERISTICS:
Population: 30 participants were dosed based on initial screening. Then 3 of the 30 participants were removed after receiving one dose because they failed inclusion/exclusion criteria leaving 27 participants to continue in the study. The baseline demographics were assessed based on the total initial enrolled number of participants (30). All 30 participants were exposed to study drug so they were in the safety population, but not all were in the efficacy as they did not continue in the study per protocol.
Groups:
- F-652 and Systemic Coritcosteroids: Subjects will be dosed once a week for four weeks with Recombinant Human Interleukin-22 IgG2-Fc (F-652). Dosing will be concurrent with systemic corticosteroids.
  Recombinant Human Interleukin-22 IgG2-Fc (F-652): IV infusion of reconstitution lyophilized F-652.
  Systemic Corticosteroids: Prednisone (or equivalent) was at the time of the onset of clinical symptoms consistent with GI and/or liver aGVHD, as per the standard of care. Prednisone (or equivalent) will be given at a dose of 2 mg/kg/day and tapered as needed.
Arm/Group | F-652 and Systemic Coritcosteroids
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.1 (15.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 16
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 24
  Black or African American | 3
  Asian | 2
  Other | 1
Region of Enrollment [Number; unit: participants]
  United States | 30
Weight [Mean (Standard Deviation); unit: kg] | 74.47 (20.457)
Height [Mean (Standard Deviation); unit: cm] — Population: Per CSR, only 29 subjects were analyzed. One subject, site inadvertently did not collect the height.
  cm
    number analyzed (Participants) | 29
    (all) | 167.73 (10.753)

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants With Lower Gastrointestinal Acute Graft-Versus-Host-Disease Treatment Response Rate on Day 28
Description: The number of participants with lower Gastrointestinal Acute Graft-Versus-Host-Disease treatment response rate on Day 28.
Time Frame: 28 days after first treatment of F-652
Population: 30 participants were dosed based on initial screening. Then 3 of the 30 participants were removed after receiving one dose because they failed inclusion/exclusion criteria leaving 27 participants to continue in the study. All participants were exposed to study drug.
Measure: Count of Participants; unit: Participants
Groups:
- F-652 and Systemic Coritcosteroids: Subjects were dosed once a week for four weeks with Recombinant Human Interleukin-22 IgG2-Fc (F-652). Dosing were concurrent with systemic corticosteroids.
  Recombinant Human Interleukin-22 IgG2-Fc (F-652): IV infusion of reconstitution lyophilized F-652.
  Systemic Corticosteroids: Prednisone (or equivalent) was at the time of the onset of clinical symptoms consistent with GI and/or liver aGVHD, as per the standard of care. Prednisone (or equivalent) were given at a dose of 2 mg/kg/day and tapered as needed.
Arm/Group | F-652 and Systemic Coritcosteroids
Number analyzed (Participants) | 27
Participants
  Treatment Response | 19
  No Treatment Response | 8

2. Secondary Outcome: The Number of Participants With Lower GI aGVHD Treatment Response at Days 14 and 56.
Description: The number of participants with Lower GI aGVHD treatment response at days 14 and 56 categorized by complete response (CR), very good partial response (VGPR), partial response (PR), no response (NR)/stable, and progression
Time Frame: Measured at day 14 and 56 after initial dosing of F-652
Population: 30 participants were dosed based on initial screening. Then 3 of the 30 participants were removed after receiving one dose because they failed inclusion/exclusion criteria leaving 27 participants to continue in the study. All were exposed to the study drug, so they were included in the safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | F-652 and Systemic Coritcosteroids
Number analyzed (Participants) | 27
Participants
  Day 14 CR Treatment Response: number analyzed (Participants) | 21
  Day 14 CR Treatment Response | 14
  Day 14 VGPR Treatment Response: number analyzed (Participants) | 21
  Day 14 VGPR Treatment Response | 1
  Day 14 PR Treatment Response: number analyzed (Participants) | 21
  Day 14 PR Treatment Response | 4
  Day 14 No Treatment Response/Stable: number analyzed (Participants) | 21
  Day 14 No Treatment Response/Stable | 2
  Day 14 No Treatment Response/Progression: number analyzed (Participants) | 21
  Day 14 No Treatment Response/Progression | 0
  Day 56 CR Treatment Response: number analyzed (Participants) | 17
  Day 56 CR Treatment Response | 12
  Day 56 VGPR Treatment Response: number analyzed (Participants) | 17
  Day 56 VGPR Treatment Response | 2
  Day 56 PR Treatment Response: number analyzed (Participants) | 17
  Day 56 PR Treatment Response | 0
  Day 56 No Treatment Response/Stable: number analyzed (Participants) | 17
  Day 56 No Treatment Response/Stable | 1
  Day 56 No Treatment Response/Progression: number analyzed (Participants) | 17
  Day 56 No Treatment Response/Progression | 2

3. Secondary Outcome: The Number of Participants With Overall aGVHD Treatment Response at Days 14, 28, and 56.
Description: The number of participants with overall aGVHD treatment response at Days 14, 28, and 56 categorized by complete response (CR), partial response (PR), no response (NR), and progression.
Time Frame: Measured at day 14, 28 and 56 after initial dosing of F-652
Population: 30 participants were dosed based on initial screening. Then 3 of the 30 participants were removed after receiving one dose because they failed inclusion/exclusion criteria leaving 27 participants to continue with the study. All participants were exposed to the study drug, so they were included in the safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | F-652 and Systemic Coritcosteroids
Number analyzed (Participants) | 27
Participants
  Day 14 CR Treatment Response: number analyzed (Participants) | 21
  Day 14 CR Treatment Response | 14
  Day 14 VGPR Treatment Response: number analyzed (Participants) | 21
  Day 14 VGPR Treatment Response | 1
  Day 14 PR Treatment Response: number analyzed (Participants) | 21
  Day 14 PR Treatment Response | 4
  Day 14 Mixed Treatment Response: number analyzed (Participants) | 21
  Day 14 Mixed Treatment Response | 1
  Day 14 No Treatment Response/Stable: number analyzed (Participants) | 21
  Day 14 No Treatment Response/Stable | 1
  Day 14 No Treatment Response/Progression: number analyzed (Participants) | 21
  Day 14 No Treatment Response/Progression | 0
  Day 28 CR Treatment Response | 13
  Day 28 VGPR Treatment Response | 4
  Day 28 PR Treatment Response | 2
  Day 28 Mixed Treatment Response | 0
  Day 28 No Treatment Response/Stable | 5
  Day 28 No Treatment Response/Progression | 3
  Day 56 CR Treatment Response: number analyzed (Participants) | 17
  Day 56 CR Treatment Response | 12
  Day 56 VGPR Treatment Response: number analyzed (Participants) | 17
  Day 56 VGPR Treatment Response | 2
  Day 56 PR Treatment Response: number analyzed (Participants) | 17
  Day 56 PR Treatment Response | 0
  Day 56 Mixed Response Treatment Response: number analyzed (Participants) | 17
  Day 56 Mixed Response Treatment Response | 1
  Day 56 No Treatment Response/Stable: number analyzed (Participants) | 17
  Day 56 No Treatment Response/Stable | 1
  Day 56 No Treatment Response/Progression: number analyzed (Participants) | 17
  Day 56 No Treatment Response/Progression | 1

4. Secondary Outcome: The Number of Participants With Discontinuation of Immunosuppressive Medication at Day 180 and 1 Year Post Initial Dosing of F-652.
Description: The number of participants with discontinuation of immunosuppressive medication at day 180 and one year post initial dose.
Time Frame: Measured at Day 180 and 1 year after initial dosing of F-652.
Population: 30 participants were dosed based on initial screening. Then 3 of the 30 participants were removed after receiving one dose because they failed inclusion/exclusion criteria leaving 27 participants to continue with the study. All were exposed to the study drug, so they were included in the safety population. The number of participants analyzed on Day 180 and 1 year post initial dosing of study drug is 11 and 10 respectively, because these participants were not lost to follow ups.
Measure: Count of Participants; unit: Participants
Groups:
- F-652 and Systemic Coritcosteroids: Subjects were dosed once a week for four weeks with Recombinant Human Interleukin-22 IgG2-Fc (F-652). Dosing were concurrent with systemic corticosteroids.
  Recombinant Human Interleukin-22 IgG2-Fc (F-652): IV infusion of reconstitution lyophilized F-652.
  Systemic Corticosteroids: Prednisone (or equivalent) was given at the time of the onset of clinical symptoms consistent with GI and/or liver aGVHD, as per the standard of care. Prednisone (or equivalent) were given at a dose of 2 mg/kg/day and tapered as needed.
Arm/Group | F-652 and Systemic Coritcosteroids
Number analyzed (Participants) | 27
Participants
  Day 180 discontinuation of immunosuppressive medication: number analyzed (Participants) | 11
  Day 180 discontinuation of immunosuppressive medication | 11
  1 year discontinuation of immunosuppressive medication: number analyzed (Participants) | 10
  1 year discontinuation of immunosuppressive medication | 10

5. Secondary Outcome: The Number of Participants With Overall Survival at 1 Year After First Infusion of F-652.
Description: The number of participants with overall survival at 1 year after first infusion of F-652.
Time Frame: Measured 1 year after first infusion.
Population: 30 participants were dosed based on initial screening. Then 3 of the 30 participants were removed after receiving one dose because they failed inclusion/exclusion criteria leaving 27 participants to continue with the study. All were exposed to the study drug, so they were included in the safety population. On the data table below, there were 3 subjects with an event were not analyzed. 24 subjects were censored for analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | F-652 and Systemic Coritcosteroids
Number analyzed (Participants) | 27
Participants | 24

ADVERSE EVENTS:
Time Frame: AEs/SAEs were assessed from the time of screening until the end of Day 56 and all causality for mortality was assessed up to 1 year.
Description: All SAEs and AEs were those assessed as possibly, probably, or definitely related to F-652 by the study Investigator at each site. Please note: 30 participants were dosed based on initial screening, so they were included in the safety population.
Groups:
- F-652 and Systemic Coritcosteroids: Subjects were dosed once a week for four weeks with Recombinant Human Interleukin-22 IgG2-Fc (F-652). Dosing will be concurrent with systemic corticosteroids.
  Recombinant Human Interleukin-22 IgG2-Fc (F-652): IV infusion of reconstitution lyophilized F-652.
  Systemic Corticosteroids: Prednisone (or equivalent) was given at the time of the onset of clinical symptoms consistent with GI and/or liver aGVHD, as per the standard of care. Prednisone (or equivalent) were given at a dose of 2 mg/kg/day and tapered as needed.
Arm/Group | F-652 and Systemic Coritcosteroids
All-Cause Mortality (participants affected / at risk) | 4/30
Serious Adverse Events (participants affected / at risk) | 10/30
Other Adverse Events (participants affected / at risk) | 26/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | F-652 and Systemic Coritcosteroids (N=30)
enterocolitis (Gastrointestinal disorders) | 1 (1)
pyrexia (General disorders) | 1 (1)
sepsis (Infections and infestations) | 2 (3)
devise related infection (Injury, poisoning and procedural complications) | 2 (2)
klebsiella infection (Infections and infestations) | 2 (2)
streptococcal pneumonia (Infections and infestations) | 1 (1)
sinusitis (Infections and infestations) | 1 (1)
muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1)
dypsnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | F-652 and Systemic Coritcosteroids (N=30)
hypokalemia (Blood and lymphatic system disorders) | 15 (18)
hyperglycemia (Blood and lymphatic system disorders) | 11 (11)
hypomagnesemia (Blood and lymphatic system disorders) | 10 (11)
hypophosphatemia (Blood and lymphatic system disorders) | 10 (11)
hypoalbuminemia (Blood and lymphatic system disorders) | 10 (10)
hyponatremia (Blood and lymphatic system disorders) | 9 (9)
hypocalcemia (Blood and lymphatic system disorders) | 8 (8)
hyperkalemia (Blood and lymphatic system disorders) | 6 (7)
hypoglycemia (Blood and lymphatic system disorders) | 6 (7)
hypermagnesemia (Blood and lymphatic system disorders) | 5 (5)
hypertriglyceridemia (Blood and lymphatic system disorders) | 5 (5)
platelet count decreased (Blood and lymphatic system disorders) | 13 (13)
lymphocyte count decreased (Blood and lymphatic system disorders) | 11 (11)
blood alkaline phosphatase increased (Blood and lymphatic system disorders) | 10 (10)
white blood cell count decreased (Blood and lymphatic system disorders) | 9 (10)
alanine aminotransferase increased (Blood and lymphatic system disorders) | 8 (8)
blood bilirubin increased (Blood and lymphatic system disorders) | 8 (8)
neutrophil count decreased (Blood and lymphatic system disorders) | 6 (7)
aspartate aminotransferase increased (Blood and lymphatic system disorders) | 6 (6)
international normalized ratio increased (Blood and lymphatic system disorders) | 5 (5)
fatigue (General disorders) | 5 (7)
peripheral edema (General disorders) | 5 (5)
dry mouth (Gastrointestinal disorders) | 6 (6)
vomiting (Gastrointestinal disorders) | 5 (6)
dry skin (Skin and subcutaneous tissue disorders) | 7 (7)
pruritus (Skin and subcutaneous tissue disorders) | 5 (5)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (5)
anemia (Blood and lymphatic system disorders) | 12 (16)
insomnia (Psychiatric disorders) | 7 (8)
muscular weakness (Musculoskeletal and connective tissue disorders) | 9 (10)
hypertension (Vascular disorders) | 6 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-05-30): https://cdn.clinicaltrials.gov/large-docs/51/NCT02406651/Prot_000.pdf
  • Statistical Analysis Plan (2020-03-19): https://cdn.clinicaltrials.gov/large-docs/51/NCT02406651/SAP_001.pdf